CLINICAL TRIAL: NCT00730015
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial of Linaclotide Administered Orally for 12 Weeks Followed by a 4-Week Randomized Withdrawal Period in Patients With Chronic Constipation
Brief Title: Trial of Linaclotide in Patients With Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCP-103-303
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Constipation
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 145 μg linaclotide (Experimental)
  Interventions: Drug: Linaclotide
- 290 μg linaclotide (Experimental)
  Interventions: Drug: Linaclotide
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Matching Placebo — Oral, once daily
  Arms: Matching Placebo
Drug: Linaclotide — Oral, once daily
  Arms: 145 μg linaclotide; 290 μg linaclotide

SUMMARY:
The objective of this trial is to determine the efficacy and safety of linaclotide administered to patients with chronic constipation (CC). The primary efficacy parameter is the percentage of patients in each dosing group that meet the protocol definition for Complete Spontaneous Bowel Movement (CSBM) Overall Responder.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed a colonoscopy according to the AGA criteria, with no clinically significant findings
* Patient has successfully completed protocol procedures (with no clinically significant findings): physical exam, 12-lead ECG, or clinical laboratory tests
* Patient meets protocol criteria for CC: reports < 3 bowel movements per week and reports straining, lumpy or hard stools, and/or sensation of incomplete evacuation during > 25% of BMs
* Patient demonstrates continued chronic constipation through Pretreatment Period
* Patient is compliant with IVRS

Exclusion Criteria:

* Patient has history of loose or watery stools
* Patient has symptoms of or been diagnosed with Irritable Bowel Syndrome (IBS)
* Patient has a structural abnormality of the gastrointestinal (GI) tract or a disease or condition that can affect GI motility
* Patient has any protocol-excluded or clinically significant medical or surgical history that could confound the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Johnston, MD, FACP, Study Chair — Ironwood Pharmaceuticals, Inc.
Locations (101):
- United States (101):
  - Ironwood Investigational Site, Birmingham, Alabama
  - Ironwood Investigational Site, Huntsville, Alabama
  - Ironwood Investigational Site, Chandler, Arizona
  - Ironwood Investigational Site, Phoenix, Arizona
  - Ironwood Investigational Site, Tucson, Arizona
  - Ironwood Investigational Site, Tuscon, Arizona
  - Ironwood Investigational Site, Sherwood, Arkansas
  - Ironwood Investigational Site, Anaheim, California
  - Ironwood Investigational Site, Chula Vista, California
  - Ironwood Investigational Site, Encinitas, California
  - Ironwood Investigational Site, Garden Grove, California
  - Ironwood Investigational Site, Laguna Hills, California
  - Ironwood Investigational Site, Los Angeles, California
  - Ironwood Investigational Site, Orange, California
  - Ironwood Investigational Site, Sacramento, California
  - Ironwood Investigational Site, San Carlos, California
  - Ironwood Investigational Site, San Diego, California
  - Ironwood Investigational Site, Colorado Springs, Colorado
  - Ironwood Investigational Site, Bristol, Connecticut
  - Ironwood Investigational Site, Boynton Beach, Florida
  - Ironwood Investigational Site, Hollywood, Florida
  - Ironwood Investigational Site, Inverness, Florida
  - Ironwood Investigational Site, Jacksonville, Florida
  - Ironwood Investigational Site, Port Orange, Florida
  - Ironwood Investigational Site, Tampa, Florida
  - Ironwood Investigational Site, Newnan, Georgia
  - Ironwood Investigational Site, Peoria, Illinois
  - Ironwood Investigational Site, Anderson, Indiana
  - Ironwood Investigational Site, Clive, Iowa
  - Ironwood Investigational Site, Davenport, Iowa
  - Ironwood Investigational Site, Mission, Kansas
  - Ironwood Investigational Site, Overland Park, Kansas
  - Ironwood Investigational Site, Topeka, Kansas
  - Ironwood Investigational Site, Baton Rouge, Louisiana
  - Ironwood Investigational Site, Monroe, Louisiana
  - Ironwood Investigational Site, Shreveport, Louisiana
  - Ironwood Investigational Site, Annapolis, Maryland
  - Ironwood Investigational Site, Baltimore, Maryland
  - Ironwood Investigational Site, Hollywood, Maryland
  - Ironwood Investigational Site, Laurel, Maryland
  - Ironwood Investigational Site, Chesterfield, Michigan
  - Ironwood Investigational Site, Traverse City, Michigan
  - Ironwood Investigational Site, Troy, Michigan
  - Ironwood Investigational Site, Jackson, Mississippi
  - Ironwood Investigational Site, Tupelo, Mississippi
  - Ironwood Investigational Site, Jefferson City, Missouri
  - Ironwood Investigational Site, Henderson, Nevada
  - Ironwood Investigational Site, Las Vegas, Nevada
  - Ironwood Investigational Site, Cedar Knolls, New Jersey
  - Ironwood Investigational Site, Marlton, New Jersey
  - Ironwood Investigational Site, Ocean City, New Jersey
  - Ironwood Investigational Site, Albuquerque, New Mexico
  - Ironwood Investigational Site, Mineola, New York
  - Ironwood Investigational Site, Pittsford, New York
  - Ironwood Investigational Site, Asheboro, North Carolina
  - Ironwood Investigational Site, Asheville, North Carolina
  - Ironwood Investigational Site, Chapel Hill, North Carolina
  - Ironwood Investigational Site, Charlotte, North Carolina
  - Ironwood Investigational Site, Greensboro, North Carolina
  - Ironwood Investigational Site, Harrisburg, North Carolina
  - Ironwood Investigational Site, Hickory, North Carolina
  - Ironwood Investigational Site, Jacksonville, North Carolina
  - Ironwood Investigational Site, New Bern, North Carolina
  - Ironwood Investigational Site, Statesville, North Carolina
  - Ironwood Investigational Site, Summerville, North Carolina
  - Ironwood Investigational Site, Wilmington, North Carolina
  - Ironwood Investigational Site, Winston-Salem, North Carolina
  - Ironwood Investigational Site, Beachwood, Ohio
  - Ironwood Investigational Site, Cincinnati, Ohio
  - Ironwood Investigational Site, Dayton, Ohio
  - Ironwood Investigational Site, Sylvania, Ohio
  - Ironwood Investigational Site, Wadsworth, Ohio
  - Ironwood Investigational Site, Zanesville, Ohio
  - Ironwood Investigational Site, Oklahoma City, Oklahoma
  - Ironwood Investigational Site, Yukon, Oklahoma
  - Ironwood Investigational Site, Lancaster, Pennsylvania
  - Ironwood Investigational Site, Levittown, Pennsylvania
  - Ironwood Investigational Site, Pittsburgh, Pennsylvania
  - Ironwood Investigational Site, Sellersville, Pennsylvania
  - Ironwood Investigational Site, Anderson, South Carolina
  - Ironwood Investigational Site, Charleston, South Carolina
  - Ironwood Investigational Site, Simpsonville, South Carolina
  - Ironwood Investigational Site, Bristol, Tennessee
  - Ironwood Investigational Site, Chattanooga, Tennessee
  - Ironwood Investigational Site, Germantown, Tennessee
  - Ironwood Investigational Site, Kingsport, Tennessee
  - Ironwood Investigational Site, Nashville, Tennessee
  - Ironwood Investigational Site, Beaumont, Texas
  - Ironwood Investigational Site, El Paso, Texas
  - Ironwood Investigational Site, Houston, Texas
  - Ironwood Investigational Site, Irving, Texas
  - Ironwood Investigational Site, Longview, Texas
  - Ironwood Investigational Site, San Antonio, Texas
  - Ironwood Investigational Site, Ogden, Utah
  - Ironwood Investigational Site, Salt Lake City, Utah
  - Ironwood Investigational Site, Chesapeake, Virginia
  - Ironwood Investigational Site, Lynchburg, Virginia
  - Ironwood Investigational Site, Spokane, Washington
  - Ironwood Investigational Site, Vancouver, Washington
  - Ironwood Investigational Site, La Crosse, Wisconsin
  - Ironwood Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Chang L, Lembo AJ, Lavins BJ, Shiff SJ, Hao X, Chickering JG, Jia XD, Currie MG, Kurtz CB, Johnston JM. The impact of abdominal pain on global measures in patients with chronic idiopathic constipation, before and after treatment with linaclotide: a pooled analysis of two randomised, double-blind, placebo-controlled, phase 3 trials. Aliment Pharmacol Ther. 2014 Dec;40(11-12):1302-12. doi: 10.1111/apt.12985. Epub 2014 Oct 13. PMID 25312449
- [Derived] Lembo AJ, Schneier HA, Shiff SJ, Kurtz CB, MacDougall JE, Jia XD, Shao JZ, Lavins BJ, Currie MG, Fitch DA, Jeglinski BI, Eng P, Fox SM, Johnston JM. Two randomized trials of linaclotide for chronic constipation. N Engl J Med. 2011 Aug 11;365(6):527-36. doi: 10.1056/NEJMoa1010863. PMID 21830967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient Recruitment occurred from August 2008 to August 2009 at 109 U.S. study centers.
Pre-assignment Details: Patients went through a 14 to 21 day Pretreatment Period during which the patients provided qualifying bowel habit and symptoms, and rescue medicine usage information through an interactive voice response system (IVRS).
Groups:
- Linaclotide, 145μg: Linaclotide, 145μg dose, oral administration, once per day
- Linaclotide, 290μg: Linaclotide, 290μg dose, oral administration, once per day
- Placebo: Dose matched placebo, oral administration, once per day
Period: Overall Study
Arm/Group | Linaclotide, 145μg | Linaclotide, 290μg | Placebo
Started | 217 | 217 | 209
Completed | 186 | 177 | 177
Not Completed | 31 | 40 | 32
Not completed — Adverse Event | 11 | 10 | 8
Not completed — Protocol Violation | 2 | 6 | 4
Not completed — Withdrawal by Subject | 12 | 12 | 8
Not completed — Lost to Follow-up | 4 | 10 | 3
Not completed — Lack of Efficacy | 1 | 2 | 8
Not completed — Other Reason | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Linaclotide, 145μg | Linaclotide, 290μg | Placebo | Total
Number analyzed (Participants) | 217 | 217 | 209 | 643
Age Continuous [Mean (Standard Deviation); unit: years] | 47.1 (14.2) | 47.7 (14.2) | 49.3 (14.3) | 48.0 (14.3)
Age, Customized [Number; unit: Participants]
  18 years to 64 years | 190 | 190 | 181 | 561
  65 years and older | 27 | 27 | 28 | 82
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 189 | 182 | 562
  Male | 26 | 28 | 27 | 81
Region of Enrollment [Number; unit: participants]
  United States | 217 | 217 | 209 | 643

OUTCOME MEASURES:

1. Primary Outcome: Complete Spontaneous Bowel Movement (CSBM) Overall Responder
Description: A 12-week CSBM Overall Responder was defined as a patient who for at least 9 of the 12 weeks of the treatment period had a CSBM weekly frequency rate that was 3 or greater and increased by 1 or more from baseline. A CSBM was defined as a spontaneous bowel movement (SBM) that was associated with a sense of complete evacuation.
  An SBM was defined as a bowel movement (BM) that occurred in the absence of laxative, enema, or suppository use on either the calendar day of the BM or the calendar day before the BM.
Time Frame: Change from Baseline to Week 12
Population: 643 randomized patients received at least 1 dose of study drug. 642 patients were included in the Intent to Treat (ITT) Population. An observed-cases approach to missing postbaseline data was applied.
Measure: Number; unit: participants
Arm/Group | Linaclotide, 145μg | Linaclotide, 290μg | Placebo
Number analyzed (Participants) | 217 | 216 | 209
participants | 46 | 42 | 7
Statistical Analysis 1: Comparison: Linaclotide, 145μg vs Placebo; Null hypothesis: There is no difference in the proportion of 12-week CSBM overall responders between patients taking the 145-μg dose and those taking placebo. The power, adjusted for multiplicity, was expected to be at least 90% based on study NCT00402337(MCP-103-201) data; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — The p-value is still less than 0.05 after adjusting multiplicity using a serial gatekeeping multiple comparison procedure; Odds Ratio (OR) = 7.72, 95% CI 2-sided [3.41 to 17.47]
Statistical Analysis 2: Comparison: Linaclotide, 290μg vs Placebo; Null hypothesis: There is no difference in the proportion of 12-week CSBM overall responders between patients taking the 290-μg dose and those taking placebo. The power, adjusted for multiplicity, was expected to be greater than 96% based on study NCT00402337(MCP-103-201) data; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 7.21, 95% CI 2-sided [3.14 to 16.59]

2. Secondary Outcome: 12-Week Complete Spontaneous Bowel Movement (CSBM) Frequency
Description: The number of CSBMs per week.
Time Frame: Change from Baseline to Week 12
Population: 643 randomized patients received at least 1 dose of study drug. 642 patients were included in the ITT Population. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: CSBMs per Week
Arm/Group | Linaclotide, 145μg | Linaclotide, 290μg | Placebo
Number analyzed (Participants) | 217 | 216 | 209
CSBMs per Week | 1.94 (0.17) | 2.04 (0.17) | 0.45 (0.17)

3. Secondary Outcome: 12-Week Spontaneous Bowl Movement (SBM) Frequency
Description: The number of SBMs per week.
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: SBMs per Week
Arm/Group | Linaclotide, 145μg | Linaclotide, 290μg | Placebo
Number analyzed (Participants) | 217 | 216 | 209
SBMs per Week | 3.03 (0.21) | 2.98 (0.21) | 1.08 (0.22)

4. Secondary Outcome: 12-week Change in Stool Consistency
Description: The consistency of each BM was assessed using the 7-point Bristol Stool Form Scale:
  1. = separate hard lumps like nuts [difficult to pass]
  2. = sausage shaped but lumpy
  3. = like a sausage but with cracks on surface
  4. = like a sausage or snake, smooth and soft
  5. = soft blobs with clear-cut edges [passed easily]
  6. = fluffy pieces with ragged edges, a mushy stool
  7. = watery, no solid pieces [entirely liquid]
Time Frame: Change from Baseline to Week 12
Population: 643 randomized patients received at least 1 dose of study drug; 642 patients were included in the ITT Population; 101 patients with no pretreatment spontaneous bowel movements were excluded from the Stool Consistency analysis. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Linaclotide, 145μg | Linaclotide, 290μg | Placebo
Number analyzed (Participants) | 183 | 181 | 177
units on a scale | 1.85 (0.08) | 1.84 (0.08) | 0.58 (0.09)

5. Secondary Outcome: 12-week Change in Severity of Straining
Description: Severity of Straining is measured on a 5-point scale, where a value of 1 is "not at all" and a value of 5 is "an extreme amount".
Time Frame: Change from Baseline to Week 12
Population: 643 randomized patients received at least 1 dose of study drug; 642 patients were included in the ITT Population; 101 patients with no pretreatment spontaneous bowel movements were excluded from the Straining analysis. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Linaclotide, 145μg | Linaclotide, 290μg | Placebo
Number analyzed (Participants) | 183 | 181 | 177
units on a scale | -1.12 (0.05) | -1.15 (0.05) | -0.51 (0.05)

6. Secondary Outcome: 12-week Change in Abdominal Discomfort
Description: Abdominal discomfort is based on a 5-point scale where a value of l is "none" and a value of 5 is "very severe."
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Linaclotide, 145μg | Linaclotide, 290μg | Placebo
Number analyzed (Participants) | 217 | 216 | 209
units on a scale | -0.49 (0.04) | -0.44 (0.04) | -0.30 (0.04)

7. Secondary Outcome: 12-week Change in Bloating
Description: Bloating was based on a 5-point scale where a value of l is "none" and a value of 5 is "very severe".
Time Frame: Change from Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Linaclotide, 145μg | Linaclotide, 290μg | Placebo
Number analyzed (Participants) | 217 | 216 | 209
units on a scale | -0.46 (0.04) | -0.37 (0.04) | -0.22 (0.04)

8. Secondary Outcome: 12-week Change in Constipation Severity
Description: Constipation severity was based on a 5-point ordinal scale where a value of l is "none" and a value of 5 is "very severe".
Time Frame: Change from Baseline to Week 12
Population: 643 randomized patients received at least 1 dose of study drug; 642 patients were included in the ITT Population; 10 patients who dropped out prior to finishing 1 week of the trial have missing data. An observed-cases approach to missing postbaseline data was applied.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Linaclotide, 145μg | Linaclotide, 290μg | Placebo
Number analyzed (Participants) | 213 | 210 | 209
units on a scale | -0.90 (0.05) | -0.81 (0.05) | -0.27 (0.05)

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected from October 2008 through October 2009. The Treatment Period lasted 12 weeks and the Randomized Withdrawal (RW) Period started after the Treamtent Period and lasted 4 weeks.
Groups:
- Linaclotide 145μg: Linaclotide, 145μg dose, oral administration, once per day
- Linaclotide 290μg: Linaclotide, 290μg dose, oral administration, once per day
- Placebo to Linaclotide 290μg Randomized Withdrawal (RW) Period: Dose-matched placebo, oral administration, once per day or Linaclotide 290μg, oral administration, once per day.
- Linaclotide 145μg to Placebo RW Period: Linaclotide 145μg, oral administration, once per day to Dose-matched placebo, oral administration, once per day
- Linaclotide 145μg to Linaclotide 145μg RW Period: Linaclotide 145μg, oral administration, once per day to Linaclotide 145μg, oral administration, once per day
- Linaclotide 290μg to Placebo RW Period: Linaclotide 290μg, oral administration, once per day to Dose-matched placebo, oral administration, once per day
- Linaclotide 290μg to Linaclotide 290μg RW Period: Linaclotide 290μg, oral administration, once per day to Linaclotide 290μg, oral administration, once per day
Arm/Group | Linaclotide 145μg | Linaclotide 290μg | Placebo | Placebo to Linaclotide 290μg Randomized Withdrawal (RW) Period | Linaclotide 145μg to Placebo RW Period | Linaclotide 145μg to Linaclotide 145μg RW Period | Linaclotide 290μg to Placebo RW Period | Linaclotide 290μg to Linaclotide 290μg RW Period
Serious Adverse Events (participants affected / at risk) | 3/217 | 4/217 | 5/209 | 0/177 | 2/95 | 0/90 | 0/86 | 0/90
Other Adverse Events (participants affected / at risk) | 27/217 | 30/217 | 14/209 | 20/177 | 1/95 | 2/90 | 0/86 | 1/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linaclotide 145μg (N=217) | Linaclotide 290μg (N=217) | Placebo (N=209) | Placebo to Linaclotide 290μg Randomized Withdrawal (RW) Period (N=177) | Linaclotide 145μg to Placebo RW Period (N=95) | Linaclotide 145μg to Linaclotide 145μg RW Period (N=90) | Linaclotide 290μg to Placebo RW Period (N=86) | Linaclotide 290μg to Linaclotide 290μg RW Period (N=90)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parathyroid tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ectopic pregnancy (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal hemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Linaclotide 145μg (N=217) | Linaclotide 290μg (N=217) | Placebo (N=209) | Placebo to Linaclotide 290μg Randomized Withdrawal (RW) Period (N=177) | Linaclotide 145μg to Placebo RW Period (N=95) | Linaclotide 145μg to Linaclotide 145μg RW Period (N=90) | Linaclotide 290μg to Placebo RW Period (N=86) | Linaclotide 290μg to Linaclotide 290μg RW Period (N=90)
Diarrhea (Gastrointestinal disorders) | 27 | 30 | 14 | 20 | 1 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that publication cannot be made for 24 months from the date of final data lock of the study, the sponsor can review the publication prior to public release, sponsor requires a minimum 60 day review period for each publication, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request an additional delay period of 60 days in order to protect potentially patentable information.